CLINICAL TRIAL: NCT05646277
Title: Patient and Practitionners Reported Experience Measures (PREMs) Following a First Remote Orthodontic Consultation Versus a First Face-to-face Orthodontic Consultation
Brief Title: Patient Reported Experience Measures Following a First Remote Orthodontic Consultation : a Randomized Controlled Trial
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Odonto01
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Odontologic Disorders
Keywords: remote-assisted teleconsultation
MeSH Terms: conditions — Tooth Diseases | interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Test: first remote-assisted orthodontic teleconsultation
  Interventions: Other: e-Consultation
- Control: classic first consultation (face-to-face consultation)
  Interventions: Other: Consultation

INTERVENTIONS:
Other: e-Consultation — first orthodontic consultation in remote
  Groups: Test
Other: Consultation — first orthodontic consultation in face-to-face
  Groups: Control

SUMMARY:
The objective of this present randomized controlled trial was to investigate patient's and practitioner's Reported Outcomes Measures (PROMs) following a first standard face-to-face consultation versus a first orthodontic teleconsultation (video-assisted remote orthodontic consultation).

ELIGIBILITY:
Inclusion criteria :

- Patients requesting a first orthodontic consultation.

Exclusion criteria :

- children not accompanied by their legal guardian (under 18 years old).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients requesting a first orthodontic consultation in the Orthodontics Unit (Odontology, Hospital of Nice)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction between first remote-assisted orthodontic teleconsultation and classic first consultation | 8 months
  satisfaction questionnaire

SECONDARY OUTCOMES:
Overall practionner satisfaction between first remote-assisted orthodontic teleconsultation and classic first consultation | 8 months
  satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
Not scheduled